CLINICAL TRIAL: NCT06834165
Title: A Phase IV Study Evaluating the Safety and Efficacy of Neffy or Intramuscular Adrenalin in Patients With Allergic Reactions After Oral Food Challenge or Allergen Immunotherapy
Brief Title: Study Evaluating the Safety and Efficacy of Neffy or Intramuscular Adrenalin in Patients With Allergic Reactions After Oral Food Challenge or Allergen Immunotherapy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: ARS Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPI R01
Record Dates: First submitted 2025-02-18; First posted 2025-02-19 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Allergic Reactions
MeSH Terms: conditions — Hypersensitivity | interventions — Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Neffy (Active Comparator)
  Interventions: Drug: Neffy
- IM adrenaline (Active Comparator)
  Interventions: Drug: Adrenaline

INTERVENTIONS:
Drug: Neffy — Epinephrine nasal spray
  Arms: Neffy
Drug: Adrenaline — Epinephrine injection
  Arms: IM adrenaline

SUMMARY:
The study is to assess the safety of neffy or IM Adrenalin in patients who are experiencing allergic reactions after an OFC, allergen Immunotherapy (AIT), or other allergy challenge that may require epinephrine intervention.

ELIGIBILITY:
Inclusion Criteria:

* Is a patient 4 years old or greater, inclusive, who are scheduled to undergo OFC, AIT, or other relevant allergy challenge.
* Has body weight 15 kg or greater at the time of allergy challenge.
* Is willing and able to provide written informed consent prior to participating in the study. In the case of minors (<18 years old), assent can be obtained from his/her legal representative, and as much possible from the patient himself/herself.
* Patient experiences an allergic reaction that, in the opinion of the Investigator, requires treatment with epinephrine via neffy or IM Adrenalin.

Exclusion Criteria:

- Has any clinically significant medical condition that precludes treatment with epinephrine as assessed by the Investigator.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
AEs after epinephrine treatment within 2 hours | 2 hours

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Orso Health, Inc., La Jolla, California
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No